CLINICAL TRIAL: NCT06179849
Title: Artificial Intelligence-enabled Large-scale Electrocardiogram Feature Extraction and Exploring Association Between the Extracted Features and Mortality, Stroke or Various Health Outcome of Interest
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2022-1506
Record Dates: First submitted 2023-11-22; First posted 2023-12-22 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Health Status(Death, Stroke Etc)

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
* In this study, large-scale ECG data (Electrocardiogram data of all patients stored in the MUSE system by measuring standard 12-guided ECG at Severance Health Checkup at Severance Hospital from November 1, 2005 to October 31, 2022) are combined with electronic medical records, National Health Insurance Corporation data, and National Statistical Office death cause data, and the artificial intelligence algorithm is used to extract ECG features to analyze the association between death, stroke, and various health conditions, and to conduct external verification or transfer learning using public databases (e.g., UK Biobank data).
* Intended to use a web-based artificial intelligence platform to distribute computational loads generated during large-scale data processing and improve analysis accuracy and efficiency.

DETAILED DESCRIPTION:
* All patient IDs obtained from the main office are replaced by research IDs (de-identified IDs), so the actual ID is not exposed and other personal identification information (name, resident registration number) is not collected.
* Research Methods:

  1. Electrocardiogram extraction based on the criteria of subjects.
  2. Combined with extracted ECG data and National Insurance Corporation data (+ National Statistical Office cause of death data).
  3. Health out of interest (HOI) definition. Includes death, stroke, etc.
  4. The defined HOI can be extracted from Yonsei Medical Center data or from National Insurance Service data or Statistics Korea's cause of death data.
  5. Artificial intelligence model training with electrocardiogram (and clinical information diagram if necessary) as input, utilizing supervised deep learning algorithms if there is a label and unsupervised learning algorithms if there is no label.
  6. Performance evaluation for supervised learning artificial intelligence models.
  7. In the case of unsupervised learning artificial intelligence models, the association/correlation between extracted features and HOI or predictability/detectability analysis.
  8. Transfer learning can be performed by adding external verification or dielectric data to the learned model using public databases.
  9. External verification can be performed using external additional data by mounting the learned model on a web-based artificial intelligence platform.
  10. Considering large-scale data, computing workloads can be distributed using web-based artificial intelligence platforms.
  11. The analysis results can be anonymized and the analysis results can be provided to researchers through a web-based artificial intelligence platform.

ELIGIBILITY:
Inclusion Criteria:

All patients stored in the MUSE system after measuring a standard 12-guided electrocardiogram at Severance Health Checkup at Severance Hospital from November 1, 2005 to October 31, 2022

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients stored in the MUSE system after measuring a standard 12-guided electrocardiogram at Severance Health Checkup at Severance Hospital from November 1, 2005 to October 31, 2022
Sampling Method: Non-Probability Sample
Enrollment: 3000000 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with Mortality | 2 years
  Investigating the reproducibility of mortality prediction (number of patients who died regardless of any cause) from ECG data measured within 1 year before death using artificial intelligence algorithms
Number of patients with Stroke, Atrial Fibrillation, Dementia | 2 years
  Investigating the correlation of certain patterns of ECG with the possibility of stroke/Atrial Fibrillation, Dementia using artificial intelligence algorithms.

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Nam Pak, Principal Investigator — Yonsei University
Locations (1):
- Yonsei University Health System, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No